CLINICAL TRIAL: NCT03189277
Title: Clinical Characteristics, Evaluation and Management of Lung Cancer Related-pain in Northern China: a Hospital-based Cross-sectional Study
Brief Title: A Hospital Based Survey on Lung Cancer Related-pain in Northern China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Chinese PLA General Hospital (Other); Beijing Chest Hospital (Other); 307 Hospital of PLA (Other); Peking Union Medical College Hospital (Other); Beijing Chao Yang Hospital (Other); Peking University Third Hospital (Other); Peking University First Hospital (Other); The Hospital of Shunyi District Beijing (Unknown); Daxing Hospital Beijing (Unknown); Peking University Third Hospital Yanqing Hospital (Unknown); Tianjin Medical University Cancer Institute and Hospital (Other); Tianjin Medical University General Hospital (Other); Hebei Medical University Fourth Hospital (Other); Henan Cancer Hospital (Other Government); Shanxi Province Cancer Hospital (Other); Inner Mongolia People's Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); 309th Hospital of Chinese People's Liberation Army (Other)
Responsible Party: Principal Investigator, Shi Yuankai, Vice president of National Cancer Center Chinese Academy of Medical Sciences, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: CH-PT-002
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Cancer Pain; Lung Cancer
MeSH Terms: conditions — Cancer Pain; Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This cross-sectional study, utilizing two sets of questionaire designed for patients and physicians respectively, aims at the epidemiology, the clinical features, and the current status of evaluation and management of lung cancer related pain in 20 participating hospitals in Northern China.

DETAILED DESCRIPTION:
Lung malignancies have become the most common cause of mortality among patients with cancer in China. A significant proportion of lung cancer patients suffer from cancer related pain, however few studies have reported the prevalence and clinical features of such pain, especially in China.

This study is a cross-sectional survey in 20 hospitals in Northern China. We designed two separate series of questions to be answered by patients and cancer management professionals. In the patient questionaire, we collect information on the prevalence, location, intensity, impact on life of lung cancer related pain. Questions on how doctors evaluate and manage the pain are included in both the patients' and physicians' surveys. In the doctors' questionaire, we also assess current situation of cancer pain educational programs attended in medical schools and post graduation through related questions.

ELIGIBILITY:
Inclusion Criteria:

1. The patient questionaire

   * All patients (outpatient and inpatient) diagnosed with lung cancer visiting the participating hospitals on the designated day of investigation
   * Informed consent must be obtained from the participating patients
2. The physician questionaire

   * All physicians who receive lung cancer patients (outpatient and inpatient) in the participating hospitals on the designated day of investigation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a cross-sectional study of clinical features (including prevalence, intensity and impact on life) of cancer-related pain in all lung cancer patients visiting the 20 participating hospitals in northern China on the designated day in July 2017. Meanwhile, all physicians receiving lung cancer patients in these hospitals are also enrolled to evaluate current management of lung cancer related pain in northern China. The patients will be identified in both outpatient clinics and inpatient wards of the involved hospitals. Informed consent will be obtained from participating patients and those who are not willing to provide pain information of interest and refuse to sign the ICF will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of cancer-related pain in lung cancer patients in 20 hospitals in northern China | 24 hours
  the proportion of self-reported pain related to cancer affecting the enrolled lung cancer patients over the past 24 hours

IPD SHARING:
Plan to Share IPD: No